CLINICAL TRIAL: NCT01698658
Title: Clinical Data Collection for Initial Evaluation of SoftVue: a Novel Ultrasound Breast Scanner
Brief Title: Ultrasound Tomography Using SoftVue in Diagnosing Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alit Amit-Yousif, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-201; NCI-2012-01745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA022453 (NIH)
Record Dates: First submitted 2012-09-26; First posted 2012-10-03 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (SoftVue ultrasound tomography) (Experimental): Patients undergo ultrasound tomography using SoftVue. Some patients also undergo MRI of the breast.
  Interventions: Other: ultrasound tomography; Procedure: magnetic resonance imaging

INTERVENTIONS:
Other: ultrasound tomography — Undergo ultrasound tomography using SoftVue
Procedure: magnetic resonance imaging — Undergo MRI of the breast
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This clinical trial studies ultrasound tomography using SoftVue in diagnosing women with breast cancer. New diagnostic procedures, such as ultrasound tomography using SoftVue, may help find and diagnose breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the in-vivo imaging potential of SoftVue through 3-dimensional (3-D) breast imaging.

II. Acquire data for SoftVue evaluation from a cohort of 100 women receiving standard ultrasound (US) evaluation as follow-up to mammographic or palpable abnormalities and construct reflection, sound speed and attenuation images with SoftVue.

III. Evaluate the ability of SoftVue to detect dominant breast findings (i.e. major normal landmark architecture) or masses previously identified with standard diagnostic evaluation (palpation, mammography, standard US) using standard clock position and radial distance measurements from the nipple.

IV. Conduct tomographic (i.e. slice-by-slice) comparison of SoftVue with magnetic resonance imaging (MRI) findings from a subgroup of 50 patients.

OUTLINE:

Patients undergo ultrasound tomography using SoftVue. Some patients also undergo MRI of the breast.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for mammogram, breast ultrasound and/or breast MRI
* Breast size less than 22 cm diameter (ring diameter is 22cm)
* Able to read or understand and provide informed consent
* Weight < 350lbs (patient bed max weight)
* Non-pregnant and non-lactating
* No open breast or chest wounds
* No active skin infection
* No serious medical or psychiatric illnesses that would prevent informed consent

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2012-10; Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Evaluation the SoftVue system with respect to spatial resolution, contrast, sound speed resolution, and attenuation resolution | At time of procedure
  For each type of resolution, observed values will be averaged over slices for each participant and compared to milestone values. The proportion of individuals whose images meet the milestone criteria will be reported with 95% confidence intervals calculated using Wilson's method.

SECONDARY OUTCOMES:
Ability of the system to identify pathological features previously identified by other imaging modalities | At time of procedure
  The sensitivity of the SoftVue system to identify pathologic features will be estimated with 95% confidence intervals using previous imaging studies as the gold standard.
Percent agreement between SoftVue (ultrasound tomography classification) and MRI (MR Breast Imaging-Reporting and Data System [BIRADS] classification) | At time of procedure
  Will be calculated along with 95% confidence intervals.
Sound speed as a percentage measure of dense breast tissue | At time of procedure
  Compare measured sound speed values against known values for the range of tissue types imaged (e.g. fatty breasts should have average sound speeds consistent with known speeds for fatty tissue).

CONTACTS AND LOCATIONS:
Overall Officials: Alit Amit-Yousif, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States